CLINICAL TRIAL: NCT05543447
Title: DERIVO® 2heal® Study: Clinical Safety and Efficacy of the DERIVO® 2heal® Embolisation Device for Intracranial Aneurysms
Brief Title: DERIVO® 2heal® Study: Clinical Safety and Efficacy of the DERIVO® 2heal® Embolisation Device
Acronym: REheal
Status: Recruiting | Type: Observational
Sponsor: Acandis GmbH (Industry)
Responsible Party: Sponsor
Other Study IDs: REheal Version 1.3, 03.06.2025
Record Dates: First submitted 2022-09-14; First posted 2022-09-16 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2024-12

CONDITIONS: Intracranial Aneurysm; Flow Diverter
Keywords: Aneurysm; DERIVO; DERIVO 2 Heal
MeSH Terms: conditions — Intracranial Aneurysm; Aneurysm

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Device: Flow Diverter Treatment with DERIVO 2 Heal Embolisation Device — Flow diversion therapy fpr intracranial aneurysm treatment.

SUMMARY:
To analyse the clinical safety and efficacy of the DERIVO® 2heal® Embolisation Device in the standard clinical routine of flow diversion treatment with respect to the mid- and long-term clinical and angiographic outcomes.

DETAILED DESCRIPTION:
The purpose of the DERIVO® 2heal® trial is to conduct a post market clinical follow-up (PMCF) study of the use of the DERIVO® 2heal® Embolisation Device in clinical practice according to EU MDCGs guidance. The DERIVO® 2heal® Study is designed as a prospective, single-arm, multicenter, open-label, national study conducted in Germany with approximately 15 sites planned. The study aims to investigate potential residual risks associated with the use of the device and to update the clinical evaluation of the device in order to ensure the long-term safety and performance of the DERIVO® 2heal® Embolisation Device after its placing on the market. For this purpose, the DERIVO® 2heal® Study will systematically collect information on technical success, safety, and clinical success of treatment of intracranial aneurysms with DERIVO® 2heal® Embolisation Device in clinical practice.

The study duration is expected to be 36 months of enrolment and 12 months follow-up of patients. Up to 158 patients should be enroled at approx. 15 study sites in Germany.

Informed consent will be obtained from all patients prior to implantation of the DERIVO® 2heal® Embolisation Device. In exceptional cases, informed consent may be obtained after the intervention, as the study is purely data collection. It should be noted that the signed informed consent form must be obtained before recording of data in the study and prior any study-specific assessments. Informed consent process will be performed according to ICH-GCP standards. In case of emergency situations when the treatment needs to be performed immediately and informed consent cannot be given prior to the rescue treatment, the informed consent can be obtained retrospectively from the patient or patient's legal representative.

The analysis population will be consist of all patients enrolled who were treated with DERIVO® 2heal® Embolisation device or in whom an attempt of DERIVO® 2heal® Embolisation device implantation was made.

Personal data will be processed in accordance with the relevant national and international legislation and good clinical practice. Data will only be processed for the purpose of the PMCF study. Person-identifiable data will not leave the unit from which they originated, and for pseudonymized data, keys to identification numbers will be held confidentially by the responsible person. Individual patient's medical information will be recorded in the study only in pseudonymized form.

All data in this project are captured in eCRFs and stored into an electronic clinical database. Quality control and data validation procedures such as programmed automatic edit and consistency checks ensure data validity and accuracy immediately at the point of entry into this database. The database application which is used to capture electronic clinical trial data is protected from unauthorized access it is, among other features, access restricted, contains rights and roles functionalities, provides electronic authentication of data entries, maintains an electronic audit trail and provides appropriate data backup functionalities.

After data entry, study monitoring team will perform source data verification and issue monitoring queries directly in the database application.

The database will only be locked after all queries and discrepancies that may have occurred during data entry have been resolved. After database lock, data will be exported in an electronic format and transferred to the responsible biometrician for analysis. The locked database may also be used to generate subject listings and tabulations.

The results of the trial will be reported to the central Ethics Committees after the study was completed. By signing the protocol, the investigator agrees that the results of the clinical investigation may be used for publication. The investigator also agrees that is not permitted to publish any data related to the trial independent of the Sponsor.

ELIGIBILITY:
Inclusion Criteria:

* Patient to be treated with DERIVO® 2heal® Embolisation Device due to intracranial aneurysm according to IFU
* Age > 18 years
* Signed Informed Consent Form
* Patient scheduled to be treated for only one target aneurysm except multiple aneurysms located in the same target zone to be treated with one DERIVO® 2heal® Embolisation Device
* Effective use of antiplatelet medication confirmed by applicable testing method according to local standard

Exclusion Criteria:

* Previously treated aneurysms with flow diverter, stent or WEB device
* Treatment as preparation for the flow-diversion treatment does not lead to exclusion of the patient
* Patient with a ruptured aneurysm in the acute phase of bleeding
* Pre-treatment disability (mRS > 2)
* Aneurysms related to pre-existing arteriosclerotic vascular disease in the target vessel
* Contraindication against treatment with anti-platelet medication
* Female patient who is known to be pregnant or is breastfeeding or wishes to become pregnant during participation in the study
* Participating in another study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients who were selected for flow diversion therapy and will be treated with DERIVO® 2heal® Embolisation Device due to intracranial aneurysm according to clinical routine.
Sampling Method: Non-Probability Sample
Enrollment: 158 (Estimated)
Dates: Start 2022-12-15 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Primary efficacy endpoint | 6 weeks +/- 3weeks; 6months +/- 3 months; 12months +/-3months
  • Rate of complete aneurysm occlusion
Primary safety endpoint | 12month ± 3month
  * Stroke/Death Occurrence Percentage of subjects with major stroke in the territory of treated artery or neurological death post-procedure
  * Rate of device-related & procedure-related complications (e.g. ICH, in-stent stenosis, in-stent thrombosis)
Primary clinical endpoint | 6 weeks ± 3weeks; 6months ± 3 months; 12months ± 3months
  • Good Clinical outcome

SECONDARY OUTCOMES:
Secondary efficacy endpoint | Measured directly after treatment
  * Wall apposition of the flow-diverter(s) per patient as determined by the treating physician and the core-lab after treatment.
    1. Correct wall apposition in the parent vessel
    2. Gap between FD and vessel wall < 25 % of vessel diameter
    3. Gap between FD and vessel wall >25 % of vessel diameter
  * Stasis / flow changes in the aneurysm (O´Kelly Marotta Scale/Kamran grading scale)
Secondary safety endpoint | 12months ± 3months
  • Rate of participants (%) with significant parent artery stenosis (> 50%) or retreatment of the target aneurysm post-procedure

CONTACTS AND LOCATIONS:
Overall Officials: Behme Daniel, Prof., Study Director — Universitätsklinikum Magdeburg
Locations (17):
- Germany (17):
  - Universitätsklinikum Augsburg, Augsburg
  - Charité - Universitätsmedizin Berlin, Berlin
  - Klinikum Bremerhaven-Reinkenheide, Bremerhaven
  - Universitätsklinikum Köln, Cologne
  - Universitätsklinikum Carl Gustav Carus Dresden, Dresden
  - Universitätsklinikum Düsseldorf, Düsseldorf
  - Universitätsklinikum Essen, Essen
  - Krankenhaus Nordwest Frankfurt, Frankfurt am Main
  - Universitätsmedizin Halle, Halle
  - Universitätsklinikum Hamburg-Eppendorf, Hamburg
  - Westpfalz-Klinikum Kaiserslautern, Kaiserslautern
  - Universitätsklinikum Magdeburg, Magdeburg
  - Mühlenkreiskliniken | Johannes Wesling Klinikum Minden, Minden
  - Ludwig-Maximilians-Universität München, München
  - Technische Universität München, München
  - Klinikum Vest - Knappschaftskrankenhaus Recklinghausen, Recklinghausen
  - Städtisches Klinikum Solingen, Solingen